CLINICAL TRIAL: NCT01180686
Title: Comparative Effectiveness of the Multiple Thrust Impulse Instrument and the Activator IV Single Thrust Instrument in Correcting a Lumbar Spinal Manipulable Lesion and Improving Lumbar Erector Spinae Flexion-relaxation
Brief Title: Comparison of a Multiple Thrust Instrument to a Single Thrust Instrument in Treating the Low Back
Acronym: AECC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anglo-European College of Chiropractic (Other)
Responsible Party: Hugh Gemmell Principal Lecturer, Anglo-European College of Chiropractic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AECC 30610; AECC30610 (Other: Anglo-European College of Chiropractic)
Record Dates: First submitted 2010-07-30; First posted 2010-08-12 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-06

CONDITIONS: Low Back Pain
Keywords: low back pain; chiropractic; manipulation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multiple thrust Impulse instrument (Active Comparator): This instrument automatically delivers 12 thrusts at the same intensity over the joint involved.
  Interventions: Device: Multiple thrust Impulse adjusting instrument
- Single impulse Activator IV instrument (Active Comparator): This is a manual spring loaded device that delivers one thrust to the joint involved
  Interventions: Device: Activator IV single impulse instrument

INTERVENTIONS:
Device: Activator IV single impulse instrument — This is a manually operated device that delivers a single thrust into the joint involved.
  Other Names: Activator IV instrument
  Arms: Single impulse Activator IV instrument
Device: Multiple thrust Impulse adjusting instrument — A device used for delivering 12 thrusts to the involved joint of the lumbar spine.
  Other Names: Impulse adjusting instrument
  Arms: Multiple thrust Impulse instrument

SUMMARY:
The purposes of this study are to determine if there is a difference between two treatment methods of spine joints that are not moving as they should as determined by tenderness over the spine and activity of the muscles along side the spine with movement.

The hypothesis is that there will be no difference between the two types of treatment.

DETAILED DESCRIPTION:
Two specialised instruments used for treating manipulable lesions of the spine will be compared using muscle relaxation response of the erector spinae muscles and correction of the spinal manipulable lesion.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-64 years of age
* Fluent in English
* With non-specific low back pain
* No lumbar manipulation within the prior 24 hours
* Not involved in strenuous back exercise on the day preceding the study
* Have not taken pain medication for two days prior to the study

Exclusion Criteria:

* Absolute contraindications to manipulation
* Specific causes for the low back pain
* Involved in or pending litigation for low back pain
* Lumbar related leg pain

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Correction of the spinal manipulable lesion | An average of 5 minutes from the the end of first treatment
  Tests used to determine the presence of a spinal manipulable lesion (a lesion in the spine requiring manipulation) will be used post-treatment to determine of correction has been achieved.

SECONDARY OUTCOMES:
Pressure pain threshold over the spinous process | An average of 5 minutes from the end of the first treatment
  An instrument used to measure pressure in kilograms is placed over the spinous process of the vertebra involved and the level of pressure is recorded when the sensation of pressure changes to pain.
Surface EMG (electromyography) of the lumbar erector spinae flexion-relaxation response | An average of 5 minutes from the end of treatment.
  Surface electromyography will be used pre-treatment and post-treatment to determine if a change in muscle activity occurs with flexing the lumbar spine.

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Gemmell, DC, EdD, Principal Investigator — Anglo-European College of Chiropractic
Locations (1):
- Anglo-European College of Chiropractic, Bournemouth, Dorset, United Kingdom